CLINICAL TRIAL: NCT00945074
Title: Protocol- vs. Patient-Oriented TCM Practices: A RCT for IBS Symptom Management
Brief Title: Acupuncture/Moxibustion for Irritable Bowel Syndrome (IBS)
Acronym: Acu/MoxaIBS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: New York University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Joyce K. Anastasi, Principal Investigator, New York University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7833948; R01NR010730 (NIH)
Record Dates: First submitted 2009-07-21; First posted 2009-07-23 (Estimated); Last update posted 2016-09-22 (Estimated); Status verified 2016-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: Acupuncture; Moxibustion; Traditional Chinese Medicine; Complementary Medicine; Irritable Bowel Syndrome; IBS
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Moxibustion

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Condition 1 (Experimental): Condition 1:
  Subjects receive Standard Acu/Moxa (fixed protocol)
  Interventions: Other: Standard Acupuncture/Moxibustion (fixed protocol)
- Condition 2: Individualized Acupuncture/Moxibustion (Experimental): Condition 2:
  Subjects receive Individualized Acupuncture/Moxibustion (patient-oriented, based on traditional Chinese medicine diagnosis).
  Interventions: Other: Individualized Acupuncture/Moxibustion
- Condition 3: Control (Sham Comparator): Condition 3:
  Subjects receive Sham Acupuncture/Placebo Moxibustion (control group)
  Interventions: Other: Sham/Placebo Acupuncture/Moxibustion

INTERVENTIONS:
Other: Standard Acupuncture/Moxibustion (fixed protocol) — Acupuncture/Moxibustion
  Arms: Condition 1
Other: Individualized Acupuncture/Moxibustion — Individualized Tailored Acupuncture/Moxibustion Protocol based on TCM Diagnosis
  Arms: Condition 2: Individualized Acupuncture/Moxibustion
Other: Sham/Placebo Acupuncture/Moxibustion — Sham/Placebo Acupuncture/Moxibustion Protocol: Not-Active
  Arms: Condition 3: Control

SUMMARY:
The objective of this study is to test the efficacy of a symptom management treatment strategy, namely, Acupuncture/Moxibustion (Acu/Moxa) to improve the symptoms associated with Irritable Bowel Syndrome (IBS) in persons between the ages of 18 to 70 years.

IBS has been defined as abdominal pain or discomfort in the mid or lower gastrointestinal (GI) tract, associated with defecation or a change in bowel patterns and with features of disordered defecation. Current therapies include dietary modification, psychotherapy and pharmacological therapies. Traditional eastern approaches offer a therapeutic approach to symptom management that is subtle, holistic and holds promise as an intervention for IBS.

This study will enroll 171 men and women experiencing IBS with diarrhea (IBS-D) defined by the ROME III criteria. Subjects will be randomized (by chance) to one of three experimental intervention conditions: Condition 1,subjects receive Standard Acu/Moxa; Condition 2, subjects receive Individualized Acu/Moxa and Condition 3, subjects receive Sham Acupuncture/Placebo Moxibustion(control group).

Subjects will attend a screening/intake session followed by two treatment sessions per week for 4 weeks, one treatment session per week for 4 weeks, and 2 non-treatment follow-up sessions at weeks 12 and 24. All subjects will be assessed by a diagnostic acupuncturist (blinded to treatment assignments), receive interventions appropriate to their condition assignment by treating acupuncturists, be administered the same instruments, and submit their symptom diaries for data entry and analysis. All subjects will complete a prospective symptom diary for the duration of the study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18 to 70 years of age who have a prior diagnosis of IBS (6 months or greater)
* Verification/documentation of subject's diagnosis of IBS (ROME III criteria).
* Subjects must be experiencing recurrent abdominal pain/discomfort with two or more of the following, as described in the Rome III criteria: (1) Improvement with defecation; and/or (2) Onset associated with a change in frequency of stool; and/or (3) Onset associated with a change in form (appearance) of stool.
* Four-week prospective daily symptom diary must show: IBS with diarrhea IBS-D), defined by ROME III
* Subjects agree to complete symptom diaries and return completed diaries at all sessions.
* Women of childbearing age must agree to use an acceptable method of contraception.
* Subjects may be on antidepressants(on stable regimen for at least 6 months)

Exclusion Criteria:

* Individuals who have IBS-Mixed, IBS-Unspecified or IBS-Constipation
* Individuals who have a history of co-existing gastrointestinal, and/or gynecological, and/or urologic pathology (eg., colon cancer, colitis, Crohn's, celiac, endometriosis, prostate cancer) or lactose intolerance
* Individuals experiencing alarm symptoms according to Rome III
* Abdominal surgery, with the exception of uncomplicated removal of the appendix, uterus, or gallbladder more than 6 months prior to study entry.
* Individuals who are currently taking the following medications more than 3 days a week: antibiotics, narcotics, cholestyramine, colchicine, iron supplements, antispasmotics, benzodiazepines
* Individuals currently receiving other types of complementary therapies such as herbs, massage, reiki etc.;Individuals receiving behavioral therapies for IBS; Individuals receiving physical therapy for pelvic pain
* Pregnant women.
* Individuals with an acute medical condition, i.e., pneumonia and/or conditions that requiring acute medical attention.
* Individuals with asthma or smoke allergy
* Individuals receiving acupuncture currently and less than 6 months prior to enrollment and/or history of receiving moxibustion
* Individuals with plans for travel, lifestyle change, or other activity that would preclude attending the planned study sessions or recording daily dietary information.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Estimated)
Dates: Start 2009-07; Primary Completion 2017-04 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Patient-rated abdominal pain/discomfort and IBS-Secondary symptom rating: intestinal gas, bloating and stool consistency | Six months

SECONDARY OUTCOMES:
Global improvement (CGIS) | Six months
Quality of life (IBS-QOL & SF-36) | Six months
Psychological distress (SCL-90) | Six months

CONTACTS AND LOCATIONS:
Overall Officials: Joyce K Anastasi, PhD, DrNP, FAAN, LAc, Principal Investigator — New York University
Locations (1):
- New York University, Division of Special Studies in Symptom Management, New York, New York, United States